CLINICAL TRIAL: NCT04728867
Title: Comparison of Textbook Versus 3D Animation Versus Cadaveric Training Video in Teaching Laparoscopic Rectal Surgery: A Prospective Randomized Clinical Trial From Tertiary Care Center
Brief Title: Comparison of Textbook Versus 3D Animation Versus Cadaveric Training Video in Teaching Laparoscopic Rectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Mehmet Ayhan Kuzu, Prof. Dr., Ankara University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: I3-73-19
Record Dates: First submitted 2021-01-18; First posted 2021-01-28 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Educational Problems

STUDY DESIGN:
Intervention Model Description: prospective, randomized, blinded study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surgical textbook (Active Comparator): Volunteers in four groups were given 4 weeks to review their educational material at least two times. For this group, this will be a textbook chapter explaining the details for laparoscopic rectal surgery.
  Interventions: Other: to compare the educational effectiveness of various educational tools
- 3D animation (Active Comparator): Volunteers in four groups were given 4 weeks to review their educational material at least two times. For this group, this will be an educational animation video showing laparoscopic rectal surgery.
  Interventions: Other: to compare the educational effectiveness of various educational tools
- Cadaveric video (Active Comparator): Volunteers in four groups were given 4 weeks to review their educational material at least two times. For this group, this will be an educational cadaveric dissection video showing laparoscopic rectal surgery.
  Interventions: Other: to compare the educational effectiveness of various educational tools
- Both 3D animation + cadaveric video (Active Comparator): Volunteers in four groups were given 4 weeks to review their educational material at least two times. For this group, this will be both animation and educational cadaveric dissection video showing laparoscopic rectal surgery.
  Interventions: Other: to compare the educational effectiveness of various educational tools

INTERVENTIONS:
Other: to compare the educational effectiveness of various educational tools — This prospective, randomized, blinded study is designed to compare the educational effectiveness of various educational tools including the surgical textbook, animation, and cadaveric videos in laparoscopic rectal surgery among board-certificated surgeons.

SUMMARY:
Digital 3D animation and cadaveric videos have been increasingly used in surgical education and provide tremendous opportunity to develop new surgical educational tools, particularly during this Coronavirus-19 pandemic period.

This prospective, randomized, blinded study is designed to compare the educational effectiveness of various educational tools including the surgical textbook, animation, and cadaveric videos in laparoscopic rectal surgery among board-certificated surgeons. Initially, an electronic questionnaire assessing the knowledge about laparoscopic rectal surgery will be created and validated by the board-certificated colorectal surgeons. Exploratory and confirmatory factor analyses will be utilized to test the structure validity of the questionnaire. After the questionnaire will be sent to the graduates completing the general surgery residency program in Turkey, the volunteers will be then randomized into four groups based on the study material including a textbook, 3D animation, cadaveric video, and both 3D animation + cadaveric video. A step-by-step educational 3D animation and a cadaveric video will be prepared in order to teach the technical steps of laparoscopic rectal surgery. Volunteers in four groups were given 2 weeks to review their educational material. After the 2-weeks of the study period, the volunteers will be asked to answers the same electronic questionnaire imported in the edited live laparoscopic rectal surgery. Pre- and post-educational assessment of the questionnaire among the groups will be performed and compared.

ELIGIBILITY:
Inclusion Criteria:

* General surgeon who graduated at least 5 years ago from the residency
* General surgeon who is proficient to perform open rectal surgery
* General surgeon who was scrubbed in/assisted for laparoscopic rectal surgery
* General surgeon who is not able to perform laparoscopic rectal surgery by itself

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of rectal cancer assessment scores among the groups before and after the education | 3 months
  Rectal cancer questionnaire that assesses the knowledge about laparoscopic rectal cancer surgery. We are expecting to see improved post-educational scores (higher than 20- mean value) (rectal cancer educational questionnaire) compared to the pre-educational scores. Higher than 20 is improved and better outcomes Range: 15-25

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem Benlice, Study Director — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No